CLINICAL TRIAL: NCT02164734
Title: Efficacy of Rescue Surfactant Delivery Via Endotracheal Intubation (INSURE Technique) Versus Laryngeal Mask Airway (LMA) for Respiratory Distress Syndrome (RDS) in Preterm Neonates
Brief Title: Surfactant Via Endotracheal Tube vs. Laryngeal Mask Airway (LMA) in Preterm Neonates With Respiratory Distress Syndrome
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow to impossible recruitment during COVID-19 pandemic
Sponsor: Albany Medical College (Other)
Collaborators: University of Rochester (Other); ONY (Industry)
Responsible Party: Principal Investigator, Joaquim M.B. Pinheiro, Professor of Pediatrics, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3768
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: surfactant
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn | interventions — Intubation, Intratracheal; Laryngeal Masks; Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endotracheal intubation (Active Comparator): Endotracheal intubation for surfactant administration, following remifentanil and atropine pre-medication
  Interventions: Device: Endotracheal intubation; Drug: remifentanil
- Laryngeal mask airway (Experimental): Laryngeal mask airway insertion for surfactant administration, following atropine pre-medication
  Interventions: Device: Laryngeal mask airway

INTERVENTIONS:
Device: Endotracheal intubation
  Other Names: INSURE
  Arms: Endotracheal intubation
Device: Laryngeal mask airway
  Other Names: LMA North America
  Arms: Laryngeal mask airway
Drug: remifentanil — additional premedication in the endotracheal intubation/INSURE arm
  Arms: Endotracheal intubation

SUMMARY:
In this study, newborn babies with respiratory distress syndrome (RDS), receiving oxygen via nasal continuous airway pressure (CPAP) modalities, and needing surfactant treatment will be randomized to standard delivery of surfactant via and endotracheal tube airway (inserted after pre-medication for pain with a short-acting narcotic), or to surfactant delivery via laryngeal mask airway (LMA). The intent is to remove the airways and return babies to non-invasive CPAP support, after surfactant is given. The primary outcome measure is the rate of failure of initial surfactant therapy. Standardized failure criteria are reached: a) early, if the baby is unable to be placed back on non-invasive CPAP (i.e., needs tracheal intubation and mechanical ventilation) or, b) late, if the baby requires ventilation, retreatment with surfactant within 8 hours or more than 2 doses of surfactant.

The objective of this protocol is to reduce the need for endotracheal intubation and mechanical ventilation in preterm neonates with RDS needing rescue surfactant therapy by instilling surfactant though an LMA, while achieving comparable efficacy of surfactant treatment.

The hypothesis is that surfactant treatment through an LMA will decrease the proportion of babies with RDS who require mechanical ventilation or subsequent intubation, when compared to standard surfactant treatment following endotracheal intubation with sedation.

DETAILED DESCRIPTION:
Respiratory Distress Syndrome (RDS) due to deficiency of pulmonary surfactant is common in preterm newborns. Early treatment with surfactant improves oxygenation, reduces the need for subsequent mechanical ventilation, decreases the incidence of pulmonary air leaks and chronic lung disease and it also reduces mortality in extremely premature newborns. Optimal treatment of RDS includes surfactant therapy and avoidance of invasive mechanical ventilation by using nasal continuous positive airway pressure modes (NCPAP or NIPPV). The current standard method of surfactant delivery requires tracheal intubation and at least brief positive-pressure ventilation, as in the INSURE (Intubation-Surfactant-Extubation) approach. Because tracheal intubation causes pain and vagal-mediated physiologic instability in neonates, premedication with atropine and a narcotic is recommended. However, narcotic premedication increases respiratory depression, which may require sustained mechanical ventilation, thus contributing to the failure of INSURE. In a recent trial at our center, standard pretreatment with morphine and atropine was associated with failure of INSURE in more than 2/3 of patients. Consequently, we have recently changed our standard premedication for INSURE to the combination of atropine and remifentanil (a rapid onset, short-acting narcotic). The Laryngeal Mask Airway (LMA) is a commercially available, less invasive artificial airway that does not need to be inserted into the trachea; it is FDA-approved for use in neonates; preliminary data suggest that it can be used for surfactant administration, which in our trial was associated with a lower failure rate than the morphine plus INSURE approach.

The main objective of this study protocol is reduce the need for endotracheal intubation and mechanical ventilation in preterm neonates with mild to moderate RDS needing rescue surfactant therapy by instilling surfactant though an LMA. A second objective is to compare the efficacy of surfactant administered via LMA versus endotracheal tube (ETT) in decreasing the severity of RDS. Additionally, we will further evaluate the safety of surfactant administration via LMA.

The primary hypothesis is that surfactant therapy delivered via LMA is not inferior to surfactant therapy delivered via transient intubation (INSURE technique) with short-acting narcotic premedication for mild to moderate RDS in preterm neonates.

This randomized controlled trial will include babies with mild-to-moderate RDS, less than 48 hours of age, with gestational age 27 0/7 to 36 6/7 weeks, treated with NCPAP (or other NIPPV modality) ≥ 5 cm H2O and FiO2 between 0.30 and 0.60 for at least 2 hours to maintain oxygen saturation by pulse oximetry (SpO2) 90-95%.

After informed consent is obtained, babies are randomly assigned (from sealed, opaque, consecutively numbered envelopes), to "ETT" or "LMA" groups. The "ETT" group is managed according to our current INSURE approach to surfactant therapy (endotracheal intubation following premedication with atropine + remifentanil), whereas the "LMA" group will be pre-medicated with atropine before LMA insertion for surfactant administration.

Both groups will receive Infasurf (3mL/kg) instilled in 2 aliquots via their respective airway, followed by PPV for at least 5 minutes. The artificial airway will be removed and the patient returned to NCPAP/NIPPV by 15 minutes, if spontaneous respirations are adequate. Indications for surfactant re-dosing and mechanical ventilation will be equivalent for both groups. Babies will continue or initiate assisted ventilation via ETT if any of the following occurs:

* Persistent apnea;
* Severe retractions;
* Inability to wean FiO2 < 60%

Criteria for re-dosing with surfactant:

1. Within 8 hours after first dose of surfactant:

   • FiO2 20% higher than the baseline FiO2, after excluding other obvious causes of respiratory insufficiency such as pneumothorax.

   If early re-dosing of surfactant is needed in patients of either group, it will be administered via ETT (i.e., LMA patients will be intubated, and will receive the dose of surfactant via ETT)
2. Beyond 8 hours of the first dose of surfactant:

   * FiO2 is ≥ 60%, or;
   * FiO2 is ≥ 30% associated with worsening clinical signs of RDS.

If late re-dosing is needed in patients of the LMA group, use of the LMA is permitted for the second dose. In the ETT group, all doses are given via the ETT.

ELIGIBILITY:
Inclusion Criteria:

* Mild-to-moderate RDS;
* Postnatal age 2 to 48 hours;
* Gestational age 27 0/7 to 36 6/7 weeks;
* Treated with nasal CPAP modalities ≥ 5 cm H2O and FiO2 between 0.30 and 0.60 for at least 2 hours to maintain SpO2 90-95%;
* Informed consent

Exclusion Criteria:

* Weight < 800 g;
* Airway anomalies;
* Pulmonary air leaks;
* Craniofacial or cardiothoracic malformations

Ages: 2 Hours to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2014-06; Primary Completion 2020-05-20 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim M Pinheiro, MD, MPH, Principal Investigator — Albany Medical College
Locations (1):
- Albany Medical Center, Albany, New York, United States

REFERENCES:
- [Derived] Gallup JA, Ndakor SM, Pezzano C, Pinheiro JMB. Randomized Trial of Surfactant Therapy via Laryngeal Mask Airway Versus Brief Tracheal Intubation in Neonates Born Preterm. J Pediatr. 2023 Mar;254:17-24.e2. doi: 10.1016/j.jpeds.2022.10.009. Epub 2022 Oct 12. PMID 36241051

RESULTS

PARTICIPANT FLOW:
Groups:
- Endotracheal Intubation: Endotracheal intubation for surfactant administration, following remifentanil and atropine pre-medication
  Endotracheal intubation
  remifentanil: additional premedication in the endotracheal intubation/INSURE arm
- Laryngeal Mask Airway: Laryngeal mask airway insertion for surfactant administration, following atropine pre-medication
  Laryngeal mask airway
Period: Overall Study
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway
Started | 42 | 51
Completed (Intention-to-treat analysis) | 42 | 51
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intention-to-treat analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway | Total
Number analyzed (Participants) | 42 | 51 | 93
Age, Continuous [Mean (Standard Deviation); unit: Gestational weeks] — Gestational age (completed weeks)
  Gestational weeks | 31.6 (2.6) | 31.7 (2.1) | 31.7 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 22 | 30 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 42 | 49 | 91
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 40 | 47 | 87
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 42 | 51 | 93
Birth weight (grams) [Mean (Standard Deviation); unit: grams] | 1848 (676) | 1926 (555) | 1891 (610)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Failing to Avoid Invasive Mechanical Ventilation
Description: Failure of surfactant therapy in avoiding invasive mechanical ventilation or clinically equivalent outcomes (FiO2 > 0.60 to maintain target SpO2, second dose of surfactant within 8 hours, or more than 2 total doses of surfactant)
Time Frame: 120 hours
Population: Analysis by intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway
Number analyzed (Participants) | 42 | 51
Participants | 12 | 10

2. Secondary Outcome: Number of Surfactant Doses
Description: Mean number of surfactant doses per patient
Time Frame: 120 hours
Measure: Mean (Standard Deviation); unit: surfactant doses
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway
Number analyzed (Participants) | 42 | 51
surfactant doses | 1.6 (0.7) | 1.6 (0.8)

3. Secondary Outcome: Days on Any Respiratory Support
Description: Days on any respiratory support (i.e., other than breathing room air)
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway
Number analyzed (Participants) | 42 | 51
days | 9 [6 to 25] | 9 [6 to 21]

4. Secondary Outcome: Rate of Pneumothorax
Description: proportion of participants with pneumothorax diagnosed radiologically or by transillumination
Time Frame: 120 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway
Number analyzed (Participants) | 42 | 51
Participants | 5 | 6

5. Secondary Outcome: Rate of Bronchopulmonary Dysplasia (O2 Dependence at the Later of 28 Days of Age or 36 Weeks Postmenstrual Age)
Description: Defined as oxygen requirement at 36 weeks postmenstrual age if gestational age less than 33 weeks, or beyond 28 days of age if gestational age greater than 32 weeks
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway
Number analyzed (Participants) | 42 | 51
Participants | 2 | 1

6. Secondary Outcome: Number of Participants With Complications During Insertion of LMA or Endotracheal Tube
Description: bradycardia, airway obstruction, or cardiopulmonary resuscitation
Time Frame: 120 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway
Number analyzed (Participants) | 42 | 51
Participants | 3 | 1

7. Secondary Outcome: Mortality Rate
Description: Mortality prior to hospital discharge (any cause)
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway
Number analyzed (Participants) | 42 | 51
Participants | 1 | 0

8. Other Pre Specified Outcome: Number of Participants With Early Failure of Surfactant Therapy
Description: need of mechanical ventilation within 1 hour of surfactant therapy
Time Frame: 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway
Number analyzed (Participants) | 42 | 51
Participants | 5 | 1

ADVERSE EVENTS:
Time Frame: 3 months or NICU discharge
Description: bradycardia
Arm/Group | Endotracheal Intubation | Laryngeal Mask Airway
All-Cause Mortality (participants affected / at risk) | 1/42 | 0/51
Serious Adverse Events (participants affected / at risk) | 1/42 | 0/51
Other Adverse Events (participants affected / at risk) | 3/42 | 1/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endotracheal Intubation (N=42) | Laryngeal Mask Airway (N=51)
cardiopulmonary resuscitation (Cardiac disorders) | 1 (1) | 0 (0) — resuscitation requiring chest compressions and/or epinephrine
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endotracheal Intubation (N=42) | Laryngeal Mask Airway (N=51)
bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
airway obstruction (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
The trial was terminated before the target enrollment numbers were reached, due to slow recruitment, which became impossible soon after the onset of the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-14): https://cdn.clinicaltrials.gov/large-docs/34/NCT02164734/Prot_SAP_000.pdf